CLINICAL TRIAL: NCT00199784
Title: Hemodynamic Measurements During Cesarean Section With Spinal Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Elangesectio2005-1; EudraCT2004-004902-26/S-05049
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2009-02

CONDITIONS: Healthy
Keywords: Hemodynamic; Hypotension; Spinal; Anesthesia; Healthy pregnant women for elective cesarean section
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine

INTERVENTIONS:
Drug: Phenylephrine

SUMMARY:
The purpose of this study is to determine the effect of low dose versus standard dose spinal anesthesia with and without intravenous phenylephrine-infusion on blood pressure, cardiac output and systemic vascular resistance.

DETAILED DESCRIPTION:
Hypotension during cesarean section with spinal anesthesia is common. We compare low dose versus standard dose spinal anesthesia with and without intravenous phenylephrine-infusion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women for elective cesarean section

Exclusion Criteria

* Shorter than 160 or taller than 180 cm
* Pre-pregnant body mass index (BMI) over 32

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-06; Study Completion 2007-04

PRIMARY OUTCOMES:
Differences in cardiac output
Blood pressure
Systemic vascular resistance

SECONDARY OUTCOMES:
Nausea
Fatigue
Cardiovascular instability due to overdosing spinal anesthesia for cesarean section (CS)

CONTACTS AND LOCATIONS:
Overall Officials: Eldrid Langesæter, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Rikshospitalet-Radiumhospitalet HF, Oslo, Oslo County, Norway

REFERENCES:
- [Result] Langesaeter E, Rosseland LA, Stubhaug A. Continuous invasive blood pressure and cardiac output monitoring during cesarean delivery: a randomized, double-blind comparison of low-dose versus high-dose spinal anesthesia with intravenous phenylephrine or placebo infusion. Anesthesiology. 2008 Nov;109(5):856-63. doi: 10.1097/ALN.0b013e31818a401f. PMID 18946298